CLINICAL TRIAL: NCT02363023
Title: Prospective Comparative Study of Different Etiologic Diagnostic Methods in Ventilator Associated Pneumonia (VAP)
Brief Title: Study of Different Etiologic Diagnostic Methods in Ventilator Associated Pneumonia (VAP)
Status: Terminated | Type: Observational
Why Stopped: Lack of resources.
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Rodrigo Miquelanti Melo, Thoracic Surgeon, Federal University of Uberlandia
Other Study IDs: VAP protocol
Record Dates: First submitted 2015-01-27; First posted 2015-02-13 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Ventilator associated pneumonia; Bronchoalveolar lavage
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — All positive cultures.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VAP suspects: Collect tracheal and pulmonary secretions. All patients (n: 72) will be submitted to endotracheal aspirate, bronchoscopic and non-bronchoscopic bronchoalveolar lavage.
  Interventions: Procedure: Collect tracheal and pulmonary secretions

INTERVENTIONS:
Procedure: Collect tracheal and pulmonary secretions — Collect tracheal and pulmonary secretions (endotracheal aspirate, bronchoscopic and non-bronchoscopic bronchoalveolar lavage)

SUMMARY:
The study is designed to evaluate sensitivity, specificity and accuracy of non-bronchoscopic bronchoalveolar lavage and endotracheal aspirate in comparison with bronchoscopic bronchoalveolar lavage (gold standard), as methods for etiologic diagnosis of ventilator associated pneumonia and their impact in morbimortality.

DETAILED DESCRIPTION:
Ventilator associated pneumonia is defined as one that occurs 48-72h after tracheal intubation, is classified into early and late and is responsible for a mortality of 24-50% to almost 70% in some studies.

The clinical suspicion of ventilator associated pneumonia is based on the finding of new or progressive pulmonary opacity associated with two or more variables such as: fever, leukocytosis or leukopenia, and purulent pulmonary secretions.

Some studies show that the etiologic diagnosis reduces spectrum of antimicrobials and bacterial resistance, reducing hospital stay and time of mechanical ventilation, as well as treatment costs. The collection of material for quantitative culture ensures greater specificity however there is no standard method.

The investigator's hypothesis is that collection of material to confirm the etiologic diagnosis of ventilator associated pneumonia, held by bronchoscopic bronchoalveolar lavage, define the etiology in a larger number of patients when compared to the endotracheal aspirate and non-bronchoscopic bronchoalveolar lavage.

The primary goal is evaluate and compare the sensitivity and specificity of noninvasive methods (endotracheal aspirate and non-bronchoscopic bronchoalveolar lavage) in comparison with invasive (bronchoscopic bronchoalveolar lavage) regarding the collection of material for etiologic diagnosis.

The secondary objectives are determine the prevalence of ventilator associated pneumonia and antimicrobial susceptibility patterns of bacteria isolated, helping to update empirical antibiotic therapy protocols.

This is a prospective comparative observational study on etiologic methods of diagnosis. All the patients, with clinical suspicion, will be submitted to collection of tracheal aspirate, bronchoscopic and non-bronchoscopic bronchoalveolar lavage. These procedures are already incorporated in the daily practice of our intensive cara unit and are routinely performed for investigation of patients with compatible framework of ventilator associated pneumonia, as availability of bronchoscopist.

Whereas an analysis of variance will be performed to compare the three interventions, with a minimum difference between the treatment means, a power of 0.95 and a significance level of 0.05, with an estimation error of 0.1, will be required a total sample of 72 patients.There will be only one group of 72 patients, in which will be held in all the three samples of the study.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 and clinical suspicion of VAP;

Exclusion Criteria:

* Age less than 18 years;
* Introduction or modification of antibiotic therapy due to associated diagnosis in the first 3 days of the start of the protocol;
* No agreement with informed consent or for any other reason, expose the desire to leave the protocol at any time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients older than 18 years admitted to the ICU of Hospital de Clínicas de Uberlândia with suspected VAP will be included in the project. from february 2015 to complete the total of 72 patients required, since provided that agree with the terms of informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy | 30 days
  Sensitivity, specificity and accuracy of noninvasive methods (endotracheal aspirate and non-bronchoscopic bronchoalveolar lavage) in comparison with invasive method (bronchoscopic bronchoalveolar lavage, considered gold standard).
  Sensitivity: number of true positive cultures obtained with each noninvasive method divided by the number of positive cultures obtained from bronchoscopic bronchoalveolar lavage;
  Specificity: number of true negative cultures obtained with each noninvasive method divided by the number of negative cultures obtained from bronchoscopic bronchoalveolar lavage;
  Accuracy: number of true positive plus true negative cultures obtained with each noninvasive method divided by the number of patients (72);

SECONDARY OUTCOMES:
Prevalence of ventilator associated pneumonia (cases / time period) | 10 months
  Number of cases of ventilator associated pneumonia divided by the number of months. We hope to reach the number of 72 patients in up to 10 months.
Antimicrobial susceptibility patterns of bacteria isolated | 72-96 hours
  All isolated bacteria will be submitted to tests for antimicrobial susceptibility and resistance pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Melo, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Rodrigo Miquelanti Melo, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
We are still collecting data.

REFERENCES:
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Kollef MH. What is ventilator-associated pneumonia and why is it important? Respir Care. 2005 Jun;50(6):714-21; discussion 721-4. PMID 15913464
- [Background] Tablan OC, Anderson LJ, Besser R, Bridges C, Hajjeh R; CDC; Healthcare Infection Control Practices Advisory Committee. Guidelines for preventing health-care--associated pneumonia, 2003: recommendations of CDC and the Healthcare Infection Control Practices Advisory Committee. MMWR Recomm Rep. 2004 Mar 26;53(RR-3):1-36. PMID 15048056
- [Background] Cook DJ, Walter SD, Cook RJ, Griffith LE, Guyatt GH, Leasa D, Jaeschke RZ, Brun-Buisson C. Incidence of and risk factors for ventilator-associated pneumonia in critically ill patients. Ann Intern Med. 1998 Sep 15;129(6):433-40. doi: 10.7326/0003-4819-129-6-199809150-00002. PMID 9735080
- [Background] Safdar N, Dezfulian C, Collard HR, Saint S. Clinical and economic consequences of ventilator-associated pneumonia: a systematic review. Crit Care Med. 2005 Oct;33(10):2184-93. doi: 10.1097/01.ccm.0000181731.53912.d9. PMID 16215368
- [Background] Rea-Neto A, Youssef NC, Tuche F, Brunkhorst F, Ranieri VM, Reinhart K, Sakr Y. Diagnosis of ventilator-associated pneumonia: a systematic review of the literature. Crit Care. 2008;12(2):R56. doi: 10.1186/cc6877. Epub 2008 Apr 21. PMID 18426596
- [Background] Bonten MJ, Bergmans DC, Stobberingh EE, van der Geest S, De Leeuw PW, van Tiel FH, Gaillard CA. Implementation of bronchoscopic techniques in the diagnosis of ventilator-associated pneumonia to reduce antibiotic use. Am J Respir Crit Care Med. 1997 Dec;156(6):1820-4. doi: 10.1164/ajrccm.156.6.9610117. PMID 9412561
- [Background] Fagon JY, Chastre J, Wolff M, Gervais C, Parer-Aubas S, Stephan F, Similowski T, Mercat A, Diehl JL, Sollet JP, Tenaillon A. Invasive and noninvasive strategies for management of suspected ventilator-associated pneumonia. A randomized trial. Ann Intern Med. 2000 Apr 18;132(8):621-30. doi: 10.7326/0003-4819-132-8-200004180-00004. PMID 10766680
- [Background] Croce MA, Fabian TC, Schurr MJ, Boscarino R, Pritchard FE, Minard G, Patton JH Jr, Kudsk KA. Using bronchoalveolar lavage to distinguish nosocomial pneumonia from systemic inflammatory response syndrome: a prospective analysis. J Trauma. 1995 Dec;39(6):1134-9; discussion 1139-40. doi: 10.1097/00005373-199512000-00022. PMID 7500408
- [Background] Leo A, Galindo-Galindo J, Folch E, Guerrero A, Bosques F, Mercado R, Arroliga AC. Comparison of bronchoscopic bronchoalveolar lavage vs blind lavage with a modified nasogastric tube in the etiologic diagnosis of ventilator-associated pneumonia. Med Intensiva. 2008 Apr;32(3):115-20. doi: 10.1016/s0210-5691(08)70921-5. PMID 18381016
- [Background] Shorr AF, Sherner JH, Jackson WL, Kollef MH. Invasive approaches to the diagnosis of ventilator-associated pneumonia: a meta-analysis. Crit Care Med. 2005 Jan;33(1):46-53. doi: 10.1097/01.ccm.0000149852.32599.31. PMID 15644647
- [Background] Canadian Critical Care Trials Group. A randomized trial of diagnostic techniques for ventilator-associated pneumonia. N Engl J Med. 2006 Dec 21;355(25):2619-30. doi: 10.1056/NEJMoa052904. PMID 17182987
- [Background] Fujitani S, Yu VL. Diagnosis of ventilator-associated pneumonia: focus on nonbronchoscopic techniques (nonbronchoscopic bronchoalveolar lavage, including mini-BAL, blinded protected specimen brush, and blinded bronchial sampling) and endotracheal aspirates. J Intensive Care Med. 2006 Jan-Feb;21(1):17-21. doi: 10.1177/0885066605283094. PMID 16698740
- [Background] Meduri GU, Chastre J. The standardization of bronchoscopic techniques for ventilator-associated pneumonia. Chest. 1992 Nov;102(5 Suppl 1):557S-564S. doi: 10.1378/chest.102.5_supplement_1.557s. No abstract available. PMID 1424930
- [Background] Baselski VS, el-Torky M, Coalson JJ, Griffin JP. The standardization of criteria for processing and interpreting laboratory specimens in patients with suspected ventilator-associated pneumonia. Chest. 1992 Nov;102(5 Suppl 1):571S-579S. doi: 10.1378/chest.102.5_supplement_1.571s. No abstract available. PMID 1424932
- [Background] Sanchez-Nieto JM, Torres A, Garcia-Cordoba F, El-Ebiary M, Carrillo A, Ruiz J, Nunez ML, Niederman M. Impact of invasive and noninvasive quantitative culture sampling on outcome of ventilator-associated pneumonia: a pilot study. Am J Respir Crit Care Med. 1998 Feb;157(2):371-6. doi: 10.1164/ajrccm.157.2.97-02039. PMID 9476845
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig LM, Lijmer JG, Moher D, Rennie D, de Vet HC; Standards for Reporting of Diagnostic Accuracy. Towards complete and accurate reporting of studies of diagnostic accuracy: the STARD initiative. Clin Radiol. 2003 Aug;58(8):575-80. doi: 10.1016/s0009-9260(03)00258-7. PMID 12887949